CLINICAL TRIAL: NCT04169308
Title: Effects of Restylane-L® Filler Injection for Non-Surgical Rhinoplasty on First Impressions and Quality of Life (FACE-Q Scale)
Brief Title: Effects of Restylane-L® Filler Injection for Non-Surgical Rhinoplasty
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DeNova Research (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Principal Investigator, Steven H. Dayan, Principal Investigator, Clinical Assistant Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RRFI-2019
Record Dates: First submitted 2019-11-12; First posted 2019-11-19 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Deformity of Nasal Cartilage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental: Restylane-L® Filler injection (Experimental)
  Interventions: Drug: Restylane-L® Filler injection

INTERVENTIONS:
Drug: Restylane-L® Filler injection — Restylane-L® Filler injection into the soft tissue of the nose

SUMMARY:
The purpose of this research is to determine the effects of Restylane-L® Filler Injection for Non-Surgical Rhinoplasty on First Impressions and Quality of Life determined by using the FACE-Q Scale.

Secondary objectives include:

To determine the efficacy of Restylane-L® Filler injection to the nose in reduction of convexity of the nasal dorsum as measured on pre/post injection 2D photographs.

To measure changes in nasal projection and rotation after injection with Restylane-L® Filler in subset of patients who underwent nasal tip augmentation.

To determine the safety of Restylane-L® Filler injection to the nose for non-surgical rhinoplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of ages 21 and above.
2. Subjects will be required not to have had previous filler injections, or other cosmetic treatments to the nose within the last 12 months.
3. Subjects that understand the purpose and aspects of the study, freely sign the consent and complete the required treatment and follow up visit.

Exclusion Criteria:

1. Males and females below age of 21.
2. Subjects who have had previous filler injections, or other cosmetic treatments to the nose within the last 12 months.
3. Subjects who are pregnant or nursing.
4. Subjects with a known allergy or sensitivity to any component of the study ingredients.
5. Any history of bleeding disorders (iatrogenic or otherwise). This includes persons who have undergone therapy with thrombolytics, anticoagulants, or inhibitors of platelet aggregation in the preceding 3 weeks.
6. Anyone taking aspirin, ibuprofen, St. John's Wort, or high doses of Vitamin E supplements in the last 3 weeks.
7. Subjects with diseases, injuries, or disabilities of the nose, including those with autoimmune disease affecting the nose, implants, and previous surgical rhinoplasty.
8. Subjects that do not understand the purpose and aspects of the study, do not sign the consent and do not complete the required treatment and follow up visit will also be excluded.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
To determine the effects of Restylane-L® Filler injection into the nose on first impressions and quality of life based on the validated questionnaires using FACE-Q scales. | 4 weeks
  We will measure changes in first impressions using a questionnaire with categories which include social skills, academic performance, dating success, occupational success, attractiveness, financial success, relationship success, and athletic skills. The 300 independent reviewers will grade each photo on a scale of 1(least favorable) to 10 (best). Evaluation of effects on quality of life will be reported through comparison of pre/post injection quality of life survey scores filled out by patients using the validated FACE-Q PRO survey measure (categories include appraisal of nasal appearance, psychological well-being, social function, and psychological distress). Maximal reported score is 4 (very satisfied) and lowest reported score is 1 (very dissatisfied).

SECONDARY OUTCOMES:
To determine the efficacy of Restylane-L® Filler injection to the nose in reduction of convexity of the nasal dorsum as measured on pre/post injection 2D photographs. | 4 weeks
  Secondary assessment of this study is to determine the efficacy of Restylane-L® filler injection into the nose as defined by the reduction of the nasal dorsal convexity to 0mm (+/- 10% of pre injection value) as measured by differences in length of a line (from pre to post injection photos) from the highest tip of the nasal dorsum to a line drawn from the Radix to the supratip region on a lateral view 2D photograph. This will be performed through calculation of changes in nasal dorsal hump convexity for all patients. All measures will be performed in triplicate and the mean of the 3 measures will be used.
To measure changes in nasal projection and rotation after injection with Restylane-L® Filler in subset of patients who underwent nasal tip augmentation. | 4 weeks
  Subgroup analysis will be performed for the patients who also underwent augmentation of the nasal tip to measure changes in projection (in mm) and rotation (in degrees) achieved from injection of filler. We will be using the Goode method for measuring nasal projection. We will be reporting the following measurements:
  Nasal projection is the perpendicular distance between the tip-defining point and a line passing through the nasion and alar crease.
  Nasal length is the distance between the nasion and the tip-defining point. The ideal Goode ratio of 0.55 to 0.60 is the perpendicular distance between the tip-defining point and a line passing through the nasion and alar crease divided by nasal length.
  Nasal tip rotation or the nasolabial angle (normal 90-120 degrees), is the angle defined by the columellar point-to-subnasale line intersecting with subnasale-to-labrale superius line.
  The mean of the 3 measurements in (mm for distance) or (degrees for rotation) will be reported.
To determine the safety of Restylane-L® Filler injection to the nose for non-surgical rhinoplasty by recording the number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 4 weeks
  The safety profile of injecting Restylane-L® into the nose will be measured by continually monitoring for AEs during the duration of the study and reporting the total number and description of events.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Dayan, MD, Principal Investigator — DeNova Research
Locations (1):
- DeNova Research, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided